CLINICAL TRIAL: NCT06582953
Title: Advancing the Evidence for HVIPs in the Southeast: Comprehensive Patient- Centered Outcomes & Stakeholder Insights
Brief Title: HVIP Outcomes and Stakeholder Insights
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00138225
Record Dates: First submitted 2024-08-11; First posted 2024-09-03 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Firearm Injury; Violence, Physical
Keywords: violence; violence intervention programs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients, family members and healthcare providers (Other): Patients that experience violent injuries or are high risk of violence between ages of 15-35 and treated at MUSC Charleston will be enrolled. The hospital violence intervention program is incorporated into regular care of patients, and they may opt to receive services from the program (TTVIP) if they qualify and opt to participate. There is no randomization or assignment. Investigators will assess outcomes of these patients and outcomes will be assessed for between group differences between those that receive services from the program and those that do not. Patient family members and healthcare providers that care for patients will be included and are exposed to the regular healthcare and services provided to patients.
  Interventions: Behavioral: Turning the Tide Violence Intervention Program (hospital violence intervention program)

INTERVENTIONS:
Behavioral: Turning the Tide Violence Intervention Program (hospital violence intervention program) — TTVIP is already integrated into the regular care of patients who are violently injured and treated at MUSC Charleston. Client advocates provide immediate support, help with communication and provide anti-retaliation messaging to victims of violence and their families, in addition to helping support their healthcare. Patients that opt to be followed for long-term wrap-around services and live in the surrounding 3-county area are supported for months (up to 1 year) after injury and provided mentorship, service referrals (i.e. education, employment, substance abuse, injury recovery, pro-social activities, housing) and mental health services.

SUMMARY:
The study's goal is to perform an evaluation of a Southeastern hospital violence intervention program (HVIP) that includes comprehensive patient outcomes, perceived benefits and opportunities for improvement of an HVIP from the perspectives of multiple stakeholders including patients, family members and healthcare providers.

DETAILED DESCRIPTION:
Evidence demonstrates that hospital violence intervention programs (HVIPs) reduce violent injury recidivism, PTSD symptoms, improve receipt of supportive services, and demonstrate cost-savings for the healthcare system. However, it is unknown if these outcomes can be replicated in under-studied communities in the Southeast (S.E.) where few HVIPs have been implemented, and other potentially valuable outcomes remain unexamined. These may include but are not limited to, improvement in patients' healthcare experiences, self-confidence, violence risk reduction, and overall recovery. In addition, multi-sector stakeholder perspectives on how HVIPs can improve or expand to better meet communities' needs are lacking in the literature. For instance, family members and loved ones are often supported by HVIP services, but little is known about how they benefit from the intervention. Also, HVIPs integrate into the healthcare team, augmenting the care provided by the clinical staff. Little is known about how healthcare teams benefit from the work of HVIPs or how the quality of care provided is influenced by these programs. These questions are imperative to informing the implementation of HVIPs and how success might be better defined through a public health lens that considers outcomes beyond violent injury recidivism for patients, families, healthcare systems, and communities.

Further, evaluating HVIPs in under-studied communities is critical to advancing the model's evidence base, especially in communities where violence intervention investment remains low. The S.E. U.S., for example, experiences a disproportionate burden of firearm homicide, but few hospitals have adopted HVIPs. S.E. trauma centers and HVIPs uniquely serve large urban and rural geographic areas that face complex racial and economic disparities yet have fewer investments in violence prevention and safety net policies and services.

Investigators propose conducting a comprehensive evaluation of an established HVIP (Turning the Tide Violence Intervention Program, TTVIP) at an academic, non-profit level 1 trauma center in Charleston, SC that serves youth and young adult victims of community and interpersonal violence in Charleston, Dorchester, and Berkeley Counties. Most patients served by the TTVIP are victims of firearm injury (>90%), reside in the cities of Charleston and North Charleston - the latter of which ranks among U.S. cities with the highest firearm assault and homicide rates - and are disproportionately young Black males from neighborhoods with high deprivation and are Medicaid funded or uninsured. This study will advance the knowledge on HVIP outcomes, implementation from the perspective of survivors, families and healthcare team members, in addition to examining the impact of an HVIP in a S.E. state that disproportionately experiences firearm violence. The study's goal is to perform an evaluation of a S.E. HVIP (TTVIP) that includes comprehensive patient outcomes, perceived benefits of HVIPs from the perspectives of multiple stakeholders, and opportunities for HVIP improvement.

Aim 1: Assess healthcare experience, supportive service utilization, violence risk, mental health outcomes, self-confidence, perceived risk of violence and re-injury among violently injured youth and young adults, including TTVIP enrolled patients and non-enrolled patients. Investigators hypothesize that individuals that experienced violent injury and enrolled in the TTVIP will report a) more positive perception of their healthcare experience, b) higher service utilization, c) lower rates of depression and PTSD, d) lower risk of violence, e) higher confidence, and f) lower rates of violent and non-violent re-injury compared to non-enrolled victims of violence. Investigators anticipate similar rates of perceived violence risk between the two groups.

Aim 2: Examine perceptions of HVIP services, benefits, and recommendations for service improvement among HVIP enrollees and their primary caregivers/loved ones.

Aim 3: Assess perceptions of HVIP services, benefits to the healthcare team and patients, and recommendations for service improvements among healthcare staff.

ELIGIBILITY:
Inclusion Criteria (patients):

* Patients ages 16-35 treated at MUSC Charleston that experience an injury due to interpersonal or community violence
* Glasgow coma score (GCS) of 15 at the time of study enrollment

Exclusion Criteria (patients):

* Lack of capacity to consent due to altered mental status (AMS) or severe untreated mental illness
* Being under arrest or incarcerated at the time of assessment for enrollment
* Non-English speaking patients
* Ages under 15, over 35

Inclusion Criteria (loved ones/caregivers):

-Loved ones (partners), caregivers and family members of patients that enroll in the study that experienced violent injuries

Exclusion Criteria (loved ones/caregivers):

* Non-English speaking
* Cognitive impairment
* Under age 16

Inclusion Criteria (Healthcare Providers):

-Healthcare team members that cared for victims of violence in the past 6 months

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Post Traumatic Stress Disorder | Victims of violence will be screened at baseline enrollment, 3 months, 6 months and 12 months after enrollment
  PTSD: PTSD Checklist for DSM-5 (PCL) The PCL-5 is a 20-item questionnaire, corresponding to the DSM-5 symptom criteria for PTSD. The self-report rating scale is 0-4 for each symptom. Rating scale descriptors are the same: Not at all, A little bit, Moderately, Quite a bit, and Extremely. They are scored 0-4. The score is totaled (0-80), with a cut-off of 33 being indicative of PTSD and higher scores indicating worse symptoms.
Self-Esteem | Victims of violence will be assessed at baseline, 3 months, 6 months and 12 months
  Self esteem will be assessed using he Rosenberg Self Esteem Scale. This is a 10-item scale with response options that indicate level of agreement (strongly agree, agree, disagree, strongly disagree) related to statements of self esteem. Responses are scored (1-4), and totaled. Higher scores indicate higher self-esteem.
Future Firearm Violence Risk | Victims of violence will be assessed at baseline, 3 months, 6 months and 12 months after enrollment.
  Future risk of firearm violence will be assessed with the SaFTEy Score (Serious fighting, Friend weapon carrying, community Environment, and firearm Threats). This is a 4 -item survey that assesses future risk of experiencing firearm violence. Each response is scored and all are totaled. Scores range 0-10, and 10 indicates high risk of future violence.
Depression | Victims of violence will be assessed at baseline enrollment, 3 months, 6 months and 12 months after enrollment.
  The PHQ-9 (patient health questionnaire) is used to assess for depression. It is a 9 item instrument that asks about depressive symptoms. Each question has a 4 response option that assesses for frequency of having symptoms, and each question is scored 0-3. The total score ranges from 0-27. 0 - 4 indicates no depression, 5-9 mild depressive symptoms, 10-14 moderate depressive symptoms, 15-19 moderately-severe depressive symptoms, and 20-27 severe depressive symptoms.
Benefits of hospital violence intervention program implementation | Healthcare providers will be assessed with baseline assessment at enrollment (1 time cross-sectional survey)
  Healthcare providers will be surveyed on perceptions of the implementation of the Turning the Tide Violence Intervention Program (TTVIP). This is not an instrument, but questions assessing the following domains will be asked in a survey: knowledge of TTVIP services, impact on communication, medical care, trauma informed care, culturally competent care, and patient outcomes. Answer options will be based on level of agreement. Results will be reported by percentage of individuals reporting the response options.
Percentage of Patients with Criminal justice system involvement | Victims of violence will be assessed at baseline enrollment, 3 months, 6 months and 12 months after enrollment
  There will not be an instrument used. Rather, subjects will be asked if they have been subject to criminal charges, arrest and incarceration. The answer options will be in a yes/no format, and the outcome will be reported by incidence (percentage of individuals indicating criminal justice system involvement).
Percentage of Patients with Adverse Social Determinants of Health | Victims of violence will be assessed at baseline, 3 months, 6 months and 12 months after enrollment
  Social Determinants of Health will be assessed with the Accountable Health Communities (AHC) Health-Related Social Needs (HRSN) Screening tool. This tool assesses social determinants of health (SDoH) and domains being assessed for this study include housing, safety, food insecurity, transportation, ability to afford basic needs, ability to pay for utilities, employment, and social support. The questions are not scored nor is a scale used, and response options are in the form of yes/no, multiple choices categories and frequencies. Results will be reported by incidence (percentage of subjects reporting the option).
Percentage of patients with perceived risk of violence | Victims of violence will be assessed at baseline enrollment, 3 months, 6 months and 12 months after enrollment.
  An instrument will not be used. The participant will be asked in a survey to indicate their level of agreement to a statement about feeling at risk of being a victim of violence. The result will be reported by the percentage of each response.
Percentage of patients experiencing a repeat injury | Victims of violence will be assessed at 3 months, 6 months and 12 months after enrollment
  An instrument will not be used. Subjects will be asked if they have experienced a repeat injury (violent or non-violent) since enrollment in the study via survey question.
Percentage of patients with recovery service needs | Victims of violence will be assessed at baseline enrollment, 3 months, 6 months and 12 months after injury. Patient loved ones/caregivers will be assessed at baseline and 3-6 months after injury.
  This will not be an instrument. Participants will be asked in a survey to indicate which services they feel like they need to recover after experiencing injury by selecting the boxes that they feel apply (services: medical/surgical, physical therapy, occupational therapy, social work, housing assistance, food assistance, transportation assistance, financial assistance, health insurance, conflict resolution, education, employment, accessing victims of crime services, legal services). Results will be reported by the percentage of individuals indicating service needs.
Percentage of patients reporting threats of violence | Victims of violence will be assessed 3 months, 6 months and 12 months after enrollment.
  This will not be assessed with an instrument. This will be assessed with a survey question asking if the patient has experienced threats of violence.
Percentage of patients reporting favorable outcomes of Violence Intervention Services | Patients enrolled in TTVIP will be assessed at the following intervals after enrollment: 3 months, 6 months and 12 months. Loved ones/caregivers will be assessed with proxy questions 3-6 months after their loved one was enrolled.
  The iMPRoVE (Measures for Providers to Victimization Experiences) is a survey that assesses the outcomes and quality of victim intervention services within the following domains: legal/justice system, medical care and coordination, mental health focused services, crisis intervention and referral services, supportive or community advocacy services, and underserved population focused services. Each question is designed to assess if the TTVIP provided services that were perceived as beneficial to the individual related to the domain. There are two question banks - one for individuals/victims, and one for proxy (caregivers, loved ones, family members). Each question has a response option (strongly agree, agree, neither agree nor disagree, disagree, strongly disagree). It is not scaled or scored, but rather each response indicates the level of agreement to the question or statement. Results will be reported by the percentage of individuals answering the options.
Percentage of Patients Reporting Favorable Quality of Health Care | Victims of violence and loved ones/caregivers will be assessed at baseline enrollment and 3 months after enrollment.
  This will not be assessed with an instrument. Questions will be administered via survey assessing the following domains of participant perception of their healthcare: communication, cultural competence, empathy, and bias. Questions will be assessed by level of agreement and reported by percentage reporting the responses.
Percentage of patients enrolled in hospital violence intervention program | Victims of violence will be asked at baseline enrollment, 3 months, 6 months and 12 months after enrollment.
  Subjects will be asked if they are enrolled in the Turning the Tide Violence Intervention Program. It will be a yes or no question, and be reported by incidence (percentage of subjects enrolled).

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Hink, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States